CLINICAL TRIAL: NCT04737447
Title: Whole Body Vibration Training in the Treatment for Children's Incontinence - a Randomized-Controlled Trial
Acronym: WBVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Alice Hoelscher, Dr. med. Alice Catherine Hoelscher, University Children's Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10642
Record Dates: First submitted 2020-12-13; First posted 2021-02-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Incontinence, Urinary
Keywords: Whole Body Vibration Training (WBVT); Incontinence in children
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial children with incontinence will be randomly assigned in two groups: an "urophysiotherapy plus WBVT" group and a control group receiving urophysiotherapy only. Statistical analysis will be randomised-controlled and prospective. Two groups will be compared:
  Group A = 20 participants treated with standardized urophysiotherapy. Group B = 20 participants treated with standardized urophysiotherapy and WBVT. According to this parameters and statistical tests will be used. Primary and secondary outcomes will be statistically described by the average (mean, median), standard deviation, frequency and percentage. The analysis will be univariant. For continuant outcomes the Student's t-Test will be used. Chi-Square Test or Fisher's Exact Test will analyze small numbers in binary or categorical outcomes.
  The level of significance (alpha) is 0.05
Masking Description: Masking is not possible because of active patient's participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Control Group) (Active Comparator): 20 participants treated with standardized urophysiotherapy twice a week, once for 45 Minutes and then for 15 Minutes. Urophysiotherapy is a well manifested and standardized therapy in the treatment für children's incontinence after the age of five years.
  Interventions: Device: Whole Body Vibration Training
- Group B (Study Group) (Active Comparator): 20 participants treated with standardized urophysiotherapy and Whole Body Vibration training (WBVT). These patients are treated with the standardized urophysiotherapy once a week and furthermore they train with WBVT twice a week for each time 15 minutes. Criteria for modifying the device utilization are based on participant's age and therapy progress. The utilized frequency of the device is individually adapted to the participant. Older patients (> ten years old) are allowed to higher frequency standards than younger participants (< 10 years old). The amplitude (0.5 mm - 2 mm) is alternated to the participant's age and height. If side effects occur (e.g. dizziness), frequency can be alternated. The intended frequency level is between 10 an 20 Hz.
  Interventions: Device: Whole Body Vibration Training

INTERVENTIONS:
Device: Whole Body Vibration Training — Galileo® Trainer is a vibration board. The movement alternating to different sides during walking correlates with the movement on the board due to variable amplitudes and frequencies. Movements of the vibration board are quickly changing and thus simulating the tilting movements of the pelvic during walking but with higher frequency. Muscles of legs and core are activated reflexively. In our study there are performed static practices and pelvic activating practices. Each physiotherapist is experienced in the technical and practical handling of the device.
  Other Names: Galileo Training

SUMMARY:
The determined study category is a prospective clinical randomized controlled study to evaluate the effect of WBVT in combination with urophysiotherapy to playfully expand the therapeutic options for children and adolescents with incontinence. This will be the first time use of WBVT for treating incontinence in children.

DETAILED DESCRIPTION:
Approximately up to 20% of children suffer from urinary incontinence. These children and frequently their families are emotionally and behaviourally affected which in turn leads to psychological distress. Urophysiotherapy became one of the first line treatments for children with urinary incontinence. Urophysiotherapy includes pelvic floor muscles training (PFMT), a treatment method not easily applicable in children. We therefore supplement the standard training with WBVT which is already evaluated in the adult population to improve the strength of the muscles of the pelvic floor. With the medical device of Galileo® children are able to train the pelvic muscles automatically and playfully.The primary objective is to investigate the effect of WBVT on children's incontinence measured by validated incontinence scores (DVISS, RUIS). The secondary objective is to evaluate the effect on the bladder function (uroflowmetry, residual urine).The primary outcome is to significantly improve incontinence symptoms by using WBVT in combination with urophysiotherapy for 9 weeks measured by incontinence scores.I nclusion criteria

* Male and Female participants 7-16 years of age
* Daytime incontinence (> 6 months)
* Written informed consent by the participant after information about the research project Exclusion criteria
* Neurogenic bladder dysfunction
* Congenital anomalies of the urinary tract
* Patients who already take part in another study concerning treating incontinence 30 days before and after participation in this study
* Patients with incontinence, who already underwent urophysiotherapy
* Medication for treating incontinence

  • Contraindications for the use of Galileo®: epilepsy, acute fractures, urolithiasis, cholecystolithaisis, after recent surgery, acute hernia, arthritis, thrombosis, rheumatic diseases, acute discopathy, patients with implants diabetes or pregnancy.
* Patients and parents without any motivation for urophysiotherapy
* Patients who neither mentally nor physically are able to pursue urophysiotherapy

In this randomized controlled trial children with incontinence will be randomly assigned in two groups: an "urophysiotherapy plus WBVT" group and a control group receiving urophysiotherapy only. The children will be treated in both groups according to a standardized protocol for 9 weeks. In addition to clinical investigations and urodynamic studies two different incontinence scores (DVISS and RUIS) will be used to determine the severity of incontinence at the time of diagnosis, at the end of the therapy (12 weeks after assessment), 24 and at 48 weeks after assessment. To determine the effect of WBVT the results will be compared using the Student's t-test and the Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants 7-16 years of age
* Daytime incontinence (> 6 months)
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* Neurogenic bladder dysfunction
* Congenital anomalies of the urinary tract
* Patients who already take part in another study concerning treating incontinence 30 days before and after participation in this study
* Patients with incontinence, who already underwent urophysiotherapy
* Medication for treating incontinence
* Contraindications for the use of Galileo®: epilepsy, acute fractures, urolithiasis, cholecystolithaisis, after recent surgery, acute hernia, arthritis, thrombosis, rheumatic diseases, acute discopathy, patients with implants diabetes or pregnancy.
* Patients and parents without any motivation for urophysiotherapy
* Patients who neither

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change of Dysfunctional Voiding and Incontinence Score (DVISS) | Change of DVISS between Baseline and Post-interventional at 12 weeks after Beginning of Intervention, 24 and 48 weeks after Intervention
  Incontinence score for children.This statistically validated functional voiding problems symptom score may provide accurate, objective and scientific bases to grade the symptoms in comparative research, diagnosis, treatment and followup of patients with wetting and functional voiding disorders. It contains 13 questions.
  The following applies:
  A child is continent when score is < 9 points and therefore responding to the therapy. Score decrease more than 30% means partial responding. Score decrease less than 30% means the failure of therapy.
Change of Revised Urinary Incontinence Scale (RUIS) | Change of RUIS between Baseline and post-interventional (12 weeks after Beginning of Intervention, 24 and 48 weeks after Intervention)
  Incontinence Score for adults.The RUIS is a short, reliable and valid five item scale that can be used to assess urinary incontinence and to monitor patient outcomes following treatment.
  The following applies:
  Incontinence is mild if scoring is less than 4, incontinence is moderate if scoring is between 4 and 8 and severe if it is more than 13.

SECONDARY OUTCOMES:
Change of Urinary flow measurements (UF) | Change of UF between Baseline and post-interventional (12 weeks after Beginning of Intervention, 24 and 48 weeks after Intervention)
  Urinary flow rate assessment is a basic noninvasive urodynamic test that is widely used to distinguish micturition problems. Key parameters are maximal flow rate (Qmax), voided volume, and flow pattern. Uroflowmetry parameters should ideally be evaluated when the voided volume is > 150 mL. The diagnostic accuracy of uroflowmetry for detecting bladder outlet obstruction varies considerably and is substantially influenced by diagnostic threshold values. Low Qmax can arise as a consequence of bladder outlet obstruction, detrusor underactivity, or an underfilled bladder.
Change of Postvoid residual urine (PVR) | Change of PVR between Baseline and post-interventional (12 weeks after Beginning of Intervention, 2 weeks after Beginning of Intervention, 24 and 48 weeks after Intervention)
  Postvoid residual urine (PVR) is the amount of urine retained in the bladder after a voluntary void and functions as a diagnostic tool. In our study, it is measured by bladder scan after urinary flow measurement to detect how much urine is left in the bladder.

CONTACTS AND LOCATIONS:
Overall Officials: Hoelscher, Principal Investigator — Consultant in Pediatric Urology
Locations (1):
- University Children's Hospital, Zurich, Switzerland